CLINICAL TRIAL: NCT04186936
Title: An Open-label, Randomized, Fasting, Two-period, Single-dose, Crossover Study to Assess Bioequivalence Between a Combination Caplet With Loperamide Hydrochloride and Simethicone (Janssen-Cilag, France), and Imodium® Express Tablets-lyophilizate (Janssen-Cilag, France) Coadministered With Espumisan® Capsule (Berlin-Chemie AG, Germany), in Healthy Volunteers
Brief Title: A Study of Combination Caplet With Loperamide Hydrochloride and Simethicone, and Imodium Express Tablets-lyophilizate Coadministered With Espumisan Capsule in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CO-161213141338-DHCT; CO-161213141338-DHCT (Other: McNeil AB)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — Loperamide; Simethicone; Espumisan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive Test Product A (single dose of 2 caplets [Combination caplet with loperamide hydrocloride [HCl] 2 milligram [mg] + simethicone 125 mg]) orally on Day 1 followed by Reference Product B (single dose of 2 Imodium Express tablets-lyophilizate [2*2 mg loperamide HCl] + 6 Espumisan capsules [6*40 mg simethicone]) orally on Day 13. A washout period of at least 7 days will be maintained between each treatment.
  Interventions: Drug: Combination Caplet with Loperamide HCl and Simethicone; Drug: Loperamide HCl; Drug: Simethicone
- Treatment Sequence BA (Experimental): Participants will receive Reference product B orally on Days 1 followed by Test product A orally on Day 13. A washout period of at least 7 days will be maintained between each treatment.
  Interventions: Drug: Combination Caplet with Loperamide HCl and Simethicone; Drug: Loperamide HCl; Drug: Simethicone

INTERVENTIONS:
Drug: Combination Caplet with Loperamide HCl and Simethicone — Participants will receive combination caplet with loperamide HCl 2 mg and simethicone 125 mg as Test product A per assigned treatment sequence.
Drug: Loperamide HCl — Participants will receive loperamide HCl 2 mg tablet-lyophilizate orally as part of Reference product B per assigned treatment sequence.
  Other Names: Imodium Express
Drug: Simethicone — Participants will receive Simethicone 40 mg capsule orally as part of Reference product B per assigned treatment sequence.
  Other Names: Espumisan

SUMMARY:
The purpose of this study is to assess bioequivalence between a Combination caplet with loperamide hydrogen chloride (HCl) 2 milligram (mg) and simethicone 125 mg, and Imodium Express tablets-lyophilizate with loperamide HCl 2 mg (co-administered with Espumisan capsules with simethicone 40 mg), with respect to the single-dose pharmacokinetics of loperamide HCl. The maximum observed concentration (Cmax), and the area under the concentration-vs.-time curve until the last measurable concentration (AUC [0-t]) will be used to assess bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 30.0 kilogram per meter (kg/m^2), inclusive, and a total body weight greater than or equal to (>=) 50.0 kilogram (kg)
* Females of childbearing potential must have a negative urine pregnancy test at the baseline visit
* Male or non-pregnant, non-lactating female agree to the contraceptive requirements (including female partner's use of a highly effective method of birth control for at least 3 months before the study, during the study and for 30 days after the last dose of investigational product)
* A personally signed and dated informed consent document before participating in any study specific procedures, indicating that the participant has been informed of all pertinent aspects of the study
* Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures specified in the protocol example: swallowing of tablets

Exclusion Criteria:

* Use of medications, prescription medication and/or over-the-counter medication including vitamins, herbal supplements, medicinal plants (example supplements containing garlic extract), and topical preparations of drugs that are systemically absorbed (example steroids and non-steroid anti-inflammatory drugs) within two weeks prior to dosing
* Use of St. John's wort (Hypericum perforatum) within 30 days prior to the first dose of study medication
* Abnormal results of laboratory and instrumental methods of examinations, including electrocardiogram (ECG)
* Females with a positive pregnancy test and/or are breast-feeding
* Females, currently using hormonal contraceptives (including use less than 2 months prior to enrollment)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  Cmax is the maximum observed concentration.
Area Under the Plasma Concentration-tme Curve From Time Zero to Time 't' (AUC[0-t]) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  AUC(0-t) is the area under the plasma concentration-time curve from time zero to time 't' (Time t is the time of the last measurable plasma concentration [Clast]).

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed measurable concentration, and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-time Curve Extrapolated from Last Measurable Concentration to Infinite Time (AUCextrap) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  AUC(extrap) is the area under the plasma concentration-time curve extrapolated from last measurable concentration to infinite time.
Time to Reach Maximum Observed Concentration (Tmax) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  Tmax is defined as time from investigational product administration to occurrence of Cmax.
Elimination Rate Constant (Lambda[z]) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  Lambda (z) is the apparent terminal elimination rate constant, estimated by linear regression using the terminal logarithmic (log)-linear phase of the log-transformed concentration versus time data.
Elimination Half-Life (t1/2) | Predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, 48, and 72 hours postdose
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Number of Participants with Adverse Events (AEs) | Up to 31 days
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Adverse Events by Severity | Up to 31 days
  The severity of AEs will be assessed by the Investigator or medically qualified individual using the following general categorical descriptors: a). Mild: Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with participant's usual function or normal everyday activities; b). Moderate: Sufficient discomfort is present to cause interference to some extent with participant's usual function or normal everyday activity; c). Severe: Extreme distress, causing significant impairment of functioning or incapacitation; interferes significantly with participants usual function; prevents normal everyday activities.
Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) | Up to 17 days
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Treatment-emergent events between administration of study drug up to 17 days that are absent before treatment or that worsened relative to pre-treatment state.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs | Up to 31 days
  Number of participants with clinically significant change from baseline in vital signs (blood pressure and heart rate) will be reported.
Number of Participants with Clinically Significant Change from Baseline in Laboratory Abnormalities | Up to 31 days
  Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count etc.), chemistry (sodium, potassium, calcium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein, glucose, creatinine and cholesterol etc.) and urine (glucose, protein, blood, ketones, nitrites, leucocyte esterase, microscopic analysis etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Anatolyevich Zacharov, Principal Investigator — McNeil AB
Locations (1):
- "Scientific and Research centre Eco-safety" Limited Liability Company, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Federal Law N 323-FZ of 21.11.2011 (as amended on 02.07.2013.) "On the basis of public health protection in the Russian Federation";
- [Background] Federal law N 61-FZ "On Circulation of Medicines" of 12.04.2010 in the edition of Federal Laws (last revised on 29.12.2015 N 389-FZ);
- [Background] Order of the RF Ministry of Health of N 266 of 19.06.2003 "On approval of clinical practice rules in the Russian Federation";
- [Background] Order of the RF Ministry of Health of N200n of 01.04.2016 "On approval of rules for Good Clinical Practice";
- [Background] Good Clinical Practice. GOST R 52379-2005 (approved by Rostechregulirovanie Order N 232-st of 27.09.2005);
- [Background] Resolution of Government of the Russian Federation N 714 of 13 September 2010 "On approval of the standard rules of the compulsory life and health insurance of the patient involved in clinical trials of the drug" (in accordance with the Governmental regulation of the Russian Federation N 393 of 18 May 2011);
- [Background] Order No 986n of Ministry of Healthcare of Russian Federation "On approval of the Regulations on the Ethics Committee" dated 29.11.2012.
- [Background] Cottrell J, Koenig K, Perfekt R, Hofmann R; Loperamide-Simethicone Acute Diarrhoea Study Team. Comparison of Two Forms of Loperamide-Simeticone and a Probiotic Yeast (Saccharomyces boulardii) in the Treatment of Acute Diarrhoea in Adults: A Randomised Non-Inferiority Clinical Trial. Drugs R D. 2015 Dec;15(4):363-73. doi: 10.1007/s40268-015-0111-y. PMID 26541878
- [Background] Hanauer SB, DuPont HL, Cooper KM, Laudadio C. Randomized, double-blind, placebo-controlled clinical trial of loperamide plus simethicone versus loperamide alone and simethicone alone in the treatment of acute diarrhea with gas-related abdominal discomfort. Curr Med Res Opin. 2007 May;23(5):1033-43. doi: 10.1185/030079907x182176. PMID 17519069
- [Background] Kaplan MA, Prior MJ, Ash RR, McKonly KI, Helzner EC, Nelson EB. Loperamide-simethicone vs loperamide alone, simethicone alone, and placebo in the treatment of acute diarrhea with gas-related abdominal discomfort. A randomized controlled trial. Arch Fam Med. 1999 May-Jun;8(3):243-8. doi: 10.1001/archfami.8.3.243. PMID 10333820
- [Background] Awouters F, Megens A, Verlinden M, Schuurkes J, Niemegeers C, Janssen PA. Loperamide. Survey of studies on mechanism of its antidiarrheal activity. Dig Dis Sci. 1993 Jun;38(6):977-95. doi: 10.1007/BF01295711. PMID 8508715
- [Background] Awouters F, Niemegeers CJ, Janssen PA. Pharmacology of antidiarrheal drugs. Annu Rev Pharmacol Toxicol. 1983;23:279-301. doi: 10.1146/annurev.pa.23.040183.001431. No abstract available. PMID 6307123
- [Background] Heykants J, Michiels M, Knaeps A, Brugmans J. Loperamide (R 18 553), a novel type of antidiarrheal agent. Part 5: the pharmacokinetics of loperamide in rats and man. Arzneimittelforschung. 1974 Oct;24(10):1649-53. No abstract available. PMID 4479779
- [Background] Heel RC, Brogden RN, Speight TM, Avery GS. Loperamide: a review of its pharmacological properties and therapeutic efficacy in diarrhoea. Drugs. 1978 Jan;15(1):33-52. doi: 10.2165/00003495-197815010-00003. PMID 342229
- [Background] Kim KA, Chung J, Jung DH, Park JY. Identification of cytochrome P450 isoforms involved in the metabolism of loperamide in human liver microsomes. Eur J Clin Pharmacol. 2004 Oct;60(8):575-81. doi: 10.1007/s00228-004-0815-3. Epub 2004 Sep 8. PMID 15365656
- [Background] Schinkel AH, Wagenaar E, Mol CA, van Deemter L. P-glycoprotein in the blood-brain barrier of mice influences the brain penetration and pharmacological activity of many drugs. J Clin Invest. 1996 Jun 1;97(11):2517-24. doi: 10.1172/JCI118699. PMID 8647944
- [Background] Cummins CL, Jacobsen W, Benet LZ. Unmasking the dynamic interplay between intestinal P-glycoprotein and CYP3A4. J Pharmacol Exp Ther. 2002 Mar;300(3):1036-45. doi: 10.1124/jpet.300.3.1036. PMID 11861813
- [Background] Mukwaya G, MacGregor T, Hoelscher D, Heming T, Legg D, Kavanaugh K, Johnson P, Sabo JP, McCallister S. Interaction of ritonavir-boosted tipranavir with loperamide does not result in loperamide-associated neurologic side effects in healthy volunteers. Antimicrob Agents Chemother. 2005 Dec;49(12):4903-10. doi: 10.1128/AAC.49.12.4903-4910.2005. PMID 16304151
- [Background] Sadeque AJ, Wandel C, He H, Shah S, Wood AJ. Increased drug delivery to the brain by P-glycoprotein inhibition. Clin Pharmacol Ther. 2000 Sep;68(3):231-7. doi: 10.1067/mcp.2000.109156. PMID 11014404
- [Background] Tayrouz Y, Ganssmann B, Ding R, Klingmann A, Aderjan R, Burhenne J, Haefeli WE, Mikus G. Ritonavir increases loperamide plasma concentrations without evidence for P-glycoprotein involvement. Clin Pharmacol Ther. 2001 Nov;70(5):405-14. doi: 10.1067/mcp.2001.119212. PMID 11719726
- [Background] Brunton L Parker K, Blumenthal D, Buxton I. Treatment of Disorders of Bowel Motility and Water Flux; Anti-Emetics; Agents Used in Biliary and Pancreatic Disease.[Book Section] // Goodman and Gilman's The Pharmacological Basis of Therapeutics. - [s.l.]: McGraw-Hill Companies Inc., 2011. - 12.
- [Background] Meier M, Steuerwald R. Review of the therapeutic use of simethicone in gastroenterology. Schweiz Z GanzheitsMedizin. 2007;19: 380-7.
- [Background] Clinical Overview. Loperamide hydrochloride. Modification of the January 2008 Company Core Data Sheet for IMODIUM® capsules, orodispersible tablets and oral solution. Document No.: EDMS-ERI-20122913. Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (December 2010).
- [Background] China Periodic Safety Update Report 01 June 2011 to 13 August 2016 ; Loperamide hydrochloride, Loperamide oxide, Loperamide/simethicone. Global Medical Safety, Janssen Research & Development, LLC, 850 Ridgeview Drive, Horsham, Pennsylvania, 19044, USA. Doc No EDMS-ERI-125782448:1.0., 28 September 2016.
- [Background] Bioequivalence report for the Modified USP in vitro defoaming test using tablets and gel capsules. Report number NG-1681985; 09 Sep 2016.
- [Background] The United States Pharmacopeial Convention. USP Monographs: Simethicone. 2000;USP29-NF 24:1518.
- [Background] Report "On experimental comparative study of toxicity of drug product Loperamide+Simethicone, tablets 2 mg+125 mg, produced by Johnson & Johnson Consumer Inc., USA (finished product manufacturer) and Janssen Cilag S.p.A., Italy (release quality control) and registered alternative drug product". // Federal State Budgetary Institution of Science "Scientific Centre of Biomedical Technologies of the Federal Medical and Biological Agency". Svetlye Gory - 2016.
- [Background] EMEA Guideline on the Investigation of Bioequivalence, January 2010, CPMP/EWP/QWP/1401/98.
- [Background] ICH Topic E 2 A Clinical Safety Data Management: Definitions and Standards for Expedited Reporting, Step 5. June 1995 CPMP/ICH/377/95.
- [Background] McNeil Study Report 15-005. An Open label, Randomized, Crossover Study to Demonstrate Bioequivalence of the Proposed Marketing Loperamide-Simethicone Caplet (batch C-826-23E) to the Currently Marketed Imodium Advanced® Caplet, and to Evaluate the Effect of Food on the Pharmacokinetics of Loperamide from the Proposed Marketing Loperamide-Simethicone Caplet. Fort Washington, PA: McNeil Consumer & Specialty Pharmaceuticals; 2006. Internal DocID: R0019405, R0024847 and R0014025.
- [Background] McNeil Study Report 98-068. Bioequivalence between Loperamide-Simethicone Caplets and Imodium® Advanced Chewable Tablets. McNeil Consumer Healthcare. Study Number CPR-154. 1999. Internal DocID: R0043738 and R0005710.
- [Background] Johnson & Johnson Study Report IMO-01. Bioequivalence between Loperamide-Simethicone Caplets and Imodium™ Plus Chewable Tables. Shandon Clinic Study Number SC00699. 2000. Internal DocID: J0041892.
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-161213141338-DHCT&attachmentIdentifier=87079b7e-b4ab-47a2-a428-d2fe06f103c1&fileName=CO-161213141338-DHCT_CSR_synopsis.pdf&versionIdentifier=